CLINICAL TRIAL: NCT00400504
Title: Hypercoagulability and Thromboembolic Risk in Patients With Malignant Disease, Evaluated by Thrombelastograph (TEG®)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: TEG-Onkologi
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2006-11-17 (Estimated); Status verified 2006-11

CONDITIONS: Cancer
Keywords: Thrombelastograph; Cancer; Thromboembolism; Hypercoagulable
MeSH Terms: conditions — Neoplasms; Thromboembolism; Thrombophilia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Patients with malignancies are at high risk of developing a thromboembolic complication and their treatment with chemo- and or radiation therapy further enhances this risk.

Conventional haemostatic tests are not suitable as a screening tool of a hypercoagulable state. A hypercoagulable profile identified with the whole blood Thrombelastograph (TEG) Analyzer parameter maximal amplitude (MA) is reported to correlate with thrombotic events in patients undergoing major non-cardial surgery and recurrent ischemic events in patients undergoing percutaneous coronary intervention.

In this study we investigate the correlation between TEG measurements and thromboembolic events in patients with newly diagnosed malignancies.

The hypotheses of this study are:

1. Patients with malignancies and hypercoagulability, defined as a TEG MA>69 mm and /or R<4 min is at increased risk of developing thromboembolic complications as compared to those with a MA<69 mm and/or a R>4 min.
2. Hypercoagulability and hence TEG R and MA values are affected by the treatment instituted in these patients (chemo and radiation therapy) rendering the patients more hypercoagulable and hence at increased risk of developing thrombotic complications.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cancer

Exclusion Criteria:

* Mamma cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Pär I Johansson, MD, Study Chair — Rigshospitalet, Denmark; Gedske Daugaard, MD, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Copenhagen, Denmark